CLINICAL TRIAL: NCT01963793
Title: Topical Aprepitant in Prurigo Patients An Exploratory Phase IIa Trial With Topically Applied Aprepitant in Patients With Prurigo
Brief Title: Topical Aprepitant in Prurigo Patients
Acronym: iTAPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0066-1019
Record Dates: First submitted 2013-09-18; First posted 2013-10-16 (Estimated); Results first posted 2021-07-16 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2021-06

CONDITIONS: Pruritus
Keywords: Pruritus
MeSH Terms: conditions — Pruritus | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (left) / aprepitant (right) (Other): placebo (on defined treatment area on left side of the body) / aprepitant (on defined treatment area on right side of the body)
  Interventions: Drug: Aprepitant; Drug: Placebo
- aprepitant (left) / placebo (right) (Other): aprepitant (on a treatment area on the left side of the body) / placebo (on a treatment area on the right side of the body)
  Interventions: Drug: Aprepitant; Drug: Placebo

INTERVENTIONS:
Drug: Aprepitant — Aprepitant gel (10 mg/g)
  Other Names: Aprepitant gel
Drug: Placebo — gel without active component
  Other Names: aprepitant gel vehicle

SUMMARY:
Topical Aprepitant in Prurigo Patients - An Exploratory Phase IIa Trial With Topically Applied Aprepitant in Patients With Prurigo

ELIGIBILITY:
Inclusion Criteria:

* Patient with Prurigo suffering from chronic pruritus
* Disease duration > six month
* Therapy refractory to at least two previous antipruritic treatments with topical, intralesional or systemic corticosteroids, or other immunosuppressants, antihistamines, antipsychotics, antidepressants, anticonvulsants and/or UV-irradiation
* Adult male or female patients, aged 18 to 80 years

Exclusion Criteria:

* Concomitant medications that are primarily metabolized through Cytochrome P450 3A4
* Applied topical antihistamines, corticosteroids or mast cell stabilizers to the skin less than 3 weeks prior to Visit 1 (Screening) or during the course of the trial
* UV-irradiation during the last 6 weeks prior to Visit 1 (Screening)
* Prescribed systemic medications are limited
* Clinically significant abnormalities in Blood analyses
* Anamnestic excessive use of alcohol or tobacco or drugs
* Presence of active tumor disease or history of malignancies within five years prior to Visit 1 (Screening)
* Known or suspected hypersensitivity to component(s) of investigational products
* Within the last 30 days or current participation in any other interventional clinical trial
* Subjects who have received treatment with any non-marketed drug substance (i.e., an agent which has not yet been made available for clinical use following registration) within the last 6 month
* Previously enrolled/randomised in this clinical trial
* In the opinion of the investigator, the subject is unlikely to comply with the Clinical Study Protocol (e.g., alcoholism, drug dependency or psychotic state)
* Females who are pregnant, of child-bearing potential and wishing to become pregnant during the trial or are breast feeding
* Females of child-bearing potential with positive pregnancy test
* Subjects (or their partner) not using an adequate method of contraception (according to national requirements, as applicable)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurer (ICI) Marcus, Prof. Dr. med., Principal Investigator — Allergie-Centrum-Charité, Charité Universitätsmedizin Berlin, Charitéplatz1, D-10117 Berlin
Locations (1):
- Allergie-Zentrum-Charité, Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Aprepitant Gel / Aprepitant Gel Vehicle: Participants were treated with aprepitant on one extremity and vehicle gel on the other 1:1 thus acting as their own intra-individual controls 10 participants: LEFT: aprepitant 10 mg/g gel , RIGHT: vehicle gel and 10 participants: LEFT: vehicle gel RIGHT: aprepitant 10 mg/g gel
Period: Overall Study
Arm/Group | Aprepitant Gel / Aprepitant Gel Vehicle
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Aprepitant Gel / Aprepitant Gel Vehicle: All 20 randomised participants were divided into two groups 1:1 10 with LEFT: aprepitant 10 mg/g gel and RIGHT: vehicle gel and 10 with LEFT: vehicle gel and RIGHT: aprepitant 10 mg/g gel
Arm/Group | Aprepitant Gel / Aprepitant Gel Vehicle
Number analyzed (Participants) | 20
Age, Continuous [Median (Standard Deviation); unit: years] | 62.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 20

OUTCOME MEASURES:

1. Primary Outcome: Pruritus by VAS (Visual Analogue Scale)
Description: At end of treatment (Day 28) participants assessed the intensity of present pruritus of each treated area on a visual analogue scale (VAS) with a score of "0" (no itch at all) to "10" (worst imaginable itch) at the two extremes on a 100 mm line.
Time Frame: At end of treatment (Day 28)
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Groups:
- Aprepitant 10 mg/g Gel: 20 participants treated with aprepitant 10mg/g gel on either left or right extremity
- Aprepitant Gel Vehicle: 20 participants were treated with vehicle gel on either left or right extremity
Arm/Group | Aprepitant 10 mg/g Gel | Aprepitant Gel Vehicle
Number analyzed (Participants) | 20 | 20
mm | 19.7 [9.5 to 29.8] | 21.2 [11.1 to 31.4]
Statistical Analysis 1: Comparison: Aprepitant 10 mg/g Gel vs Aprepitant Gel Vehicle; Test type: Superiority; p = 0.58, t-test, 2 sided; Mean Difference (Final Values) = -1.51, 95% CI 2-sided [-7.12 to 4.11]

2. Secondary Outcome: Pruritus by VAS (Visual Analogue Scale)
Description: At baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42, participants assessed the intensity of present pruritus of each treated area on a visual analogue scale (VAS) with a score of "0" (no itch at all) to "10" (worst imaginable itch) at the two extremes on a 100 mm line.
Time Frame: At baseline (Day 1), Day 14, end of treatment (Day 28), and Day 42
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Aprepitant 10 mg/g Gel | Aprepitant Gel Vehicle
Number analyzed (Participants) | 20 | 20
mm
  Day 1 (Visit 2) | 50.8 (26.6) | 58.1 (28.2)
  Day 14 (Visit 3) | 27.1 (24.2) | 28.7 (19.1)
  Day 28 (Visit 4) | 19.0 (21.0) | 21.9 (24.2)
  Day 42 (Visit 5) | 23.9 (28.2) | 24.0 (26.7)

3. Secondary Outcome: Change From Baseline in Participants' Global Assessment on Treatment Areas
Description: At baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42, participants assessed their prurigo on each treated area using the following score: 0 = no symptoms, 1 = mild, 2 = moderate, 3 = severe. The change was calculated as the value at the later time point minus the value at baseline. The change at Day 1 was therefore 0 and negative values represent a decrease in score.
Time Frame: At baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Aprepitant 10 mg/g Gel: 20 participants treated with aprepitant 10 mg/g gel on either left or right extremity
Arm/Group | Aprepitant 10 mg/g Gel | Aprepitant Gel Vehicle
Number analyzed (Participants) | 20 | 20
units on a scale
  Day 1 (Visit 2) | 0.0 (0.0) | 0.0 (0.0)
  Day 14 (Visit 3) | -0.5 (0.8) | -0.7 (0.9)
  Day 28 (Visit 4) | -0.6 (1.1) | -0.7 (1.1)
  Day 42 (Visit 5) | -0.3 (0.9) | -0.4 (0.9)

4. Secondary Outcome: Clinical Score Assessment of Crusting
Description: The (sub)investigator assessed the clinical picture at each treated area at baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42 using the following score:
  Criteria:
  Crusts
  Evaluation:
  0 = not existing
  1. = mild
  2. = moderate
  3. = severe
  The score will be an integer on the scale 0-3.
Time Frame: At baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant 10 mg/g Gel | Aprepitant Gel Vehicle
Number analyzed (Participants) | 20 | 20
units on a scale
  Day 1 (Visit 2) | 1.3 (0.9) | 1.4 (0.9)
  Day 14 (Visit 3) | 0.9 (0.9) | 1.1 (0.8)
  Day 28 (Visit 4) | 0.7 (0.8) | 1.0 (1.1)
  Day 42 (Visit 5) | 0.8 (0.8) | 0.9 (0.7)

5. Secondary Outcome: Clinical Score Assessment of Erythema
Description: The (sub)investigator will assess the clinical picture at each treated area at baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42 using the following score:
  Criteria:
  Erythema
  Evaluation:
  0 = not existing
  1. = mild
  2. = moderate
  3. = severe
  The score will be an integer on the scale 0-3.
Time Frame: At baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant 10 mg/g Gel | Aprepitant Gel Vehicle
Number analyzed (Participants) | 20 | 20
units on a scale
  Day 1 (Visit 2) | 2.0 (0.8) | 2.1 (0.8)
  Day 14 (Visit 3) | 1.8 (0.9) | 1.8 (0.9)
  Day 28 (Visit 4) | 1.5 (0.9) | 1.7 (0.9)
  Day 42 (Visit 5) | 1.5 (0.8) | 1.6 (0.7)

6. Secondary Outcome: Clinical Score Assessment of Scratch Artefacts
Description: The (sub)investigator will assess the clinical picture at each treated area at baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42 using the following score:
  Criteria:
  Scratch artefacts: Superficial damage to the skin caused by severe scratching.
  Evaluation:
  0 = not existing
  1. = mild
  2. = moderate
  3. = severe
  The score will be an integer on the scale 0-3.
Time Frame: At baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant 10 mg/g Gel | Aprepitant Gel Vehicle
Number analyzed (Participants) | 20 | 20
units on a scale
  Day 1 (Visit 2) | 1.7 (1.1) | 1.8 (1.1)
  Day 14 (Visit 3) | 1.3 (1.1) | 1.3 (1.1)
  Day 28 (Visit 4) | 1.1 (1.0) | 1.4 (1.1)
  Day 42 (Visit 5) | 1.4 (1.2) | 1.4 (1.2)

7. Secondary Outcome: Clinical Score Assessment of Infiltration
Description: The (sub)investigator will assess the clinical picture at each treated area at baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42 using the following score:
  Criteria:
  Infiltration
  Evaluation:
  0 = not existing
  1. = mild
  2. = moderate
  3. = severe
  The score will be an integer on the scale 0-3.
Time Frame: At baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant 10 mg/g Gel | Aprepitant Gel Vehicle
Number analyzed (Participants) | 20 | 20
units on a scale
  Day 1 (Visit 2) | 1.5 (1.2) | 1.5 (1.1)
  Day 14 (Visit 3) | 1.3 (1.0) | 1.4 (1.1)
  Day 28 (Visit 4) | 1.1 (0.9) | 1.3 (1.0)
  Day 42 (Visit 5) | 1.3 (0.9) | 1.5 (1.1)

8. Secondary Outcome: Transepidermal Water Loss (TEWL)
Description: The (sub)investigator will made the following clinical assessment:
  Transepidermal water loss was defined as amount of released water from skin surface in g/cm^2 per hour. The TEWL is increased in case of damage of skin barrier.
Time Frame: At baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42
Measure: Mean (Standard Deviation); unit: g/cm² per hour
Arm/Group | Aprepitant 10 mg/g Gel | Aprepitant Gel Vehicle
Number analyzed (Participants) | 20 | 20
g/cm² per hour
  Day 1 (Visit 2) | 20.6 (13.6) | 25.2 (12.8)
  Day 14 (Visit 3) | 22.7 (12.5) | 24.0 (12.5)
  Day 28 (Visit 4) | 20.0 (19.5) | 19.9 (21.3)
  Day 42 (Visit 5) | 19.4 (13.2) | 19.9 (9.7)

9. Secondary Outcome: Lesional Erythema by Mexameter
Description: The skin colour of the participants was evaluated by use of a Mexameter spectrophotometer. The instrument computed an erythema index (with a range between 0 and 999, where higher values indicate more erythema or redness) which may be used as an indication of skin properties.
  Mexameter measurements were performed at baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42 to assess stimulation of microcirculation, irritating effects, and occurring erythema.
Time Frame: At baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant 10 mg/g Gel | Aprepitant Gel Vehicle
Number analyzed (Participants) | 20 | 20
units on a scale
  Day 1 (Visit 2) | 438 (124) | 453 (107)
  Day 14 (Visit 3) | 527 (122) | 463 (119)
  Day 28 (Visit 4) | 464 (114) | 491 (147)
  Day 42 (Visit 5) | 457 (120) | 461 (144)

10. Secondary Outcome: Non-lesional Erythema by Mexameter
Description: as for outcome 9
Time Frame: At baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lateral Side of Aprepitant 10 mg/g Gel: 20 participants treated with aprepitant 10 mg/g gel on either left or right extremity
- Lateral Side of Aprepitant Gel Vehicle: 20 participants were treated with vehicle gel on either left or right extremity
Arm/Group | Lateral Side of Aprepitant 10 mg/g Gel | Lateral Side of Aprepitant Gel Vehicle
Number analyzed (Participants) | 20 | 20
units on a scale
  Day 1 (Visit 2) | 304 (151) | 300 (145)
  Day 14 (Visit 3) | 287 (84.6) | 312 (138)
  Day 28 (Visit 4) | 262 (104) | 271 (71.8)
  Day 42 (Visit 5) | 284 (79.5) | 284 (85.3)

11. Secondary Outcome: Melanin by Mexameter
Description: The skin colour of the participants was evaluated by use of a Mexameter spectrophotometer. The instrument computed a melanin index (with a range between 0 and 999, where higher values indicate more melanin) which may be used as an indication of skin properties.
  Mexameter measurements were performed at baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42 to assess stimulation of microcirculation, irritating effects, and occurring erythema.
Time Frame: At baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant 10 mg/g Gel | Aprepitant Gel Vehicle
Number analyzed (Participants) | 20 | 20
units on a scale
  Day 1 (Visit 2) | 131 (61.6) | 115 (52.4)
  Day 14 (Visit 3) | 121 (43.8) | 134 (56.8)
  Day 28 (Visit 4) | 152 (51.7) | 139 (60.3)
  Day 42 (Visit 5) | 132 (73.2) | 144 (77.5)

12. Secondary Outcome: Non-lesional Melanin by Mexameter
Description: as for outcome 11
Time Frame: At baseline (Day 1), Day 14, end of treatment (Day 28) and Day 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant 10 mg/g Gel | Aprepitant Gel Vehicle
Number analyzed (Participants) | 20 | 20
units on a scale
  Day 1 (Visit 2) | 127 (58.9) | 129 (49.0)
  Day 14 (Visit 3) | 165 (179) | 215 (224)
  Day 28 (Visit 4) | 149 (117) | 166 (170)
  Day 42 (Visit 5) | 129 (51.3) | 179 (236)

13. Secondary Outcome: Daily Assessments of Duration of Pruritus (Preceding 12 Hours)
Description: During the trial participants completed a diary twice daily, in the morning and in the evening, each covering the preceding 12 hours, which collected the number of hours with pruritus within the last 12 hours on both areas by use of a 7-point scale (<0.5 hours, 0.5-1 hours, 1-2 hours, 3-4 hours, 5-6 hours, 7-8 hours, 9-12 hours).
  Duration of pruritus was categorized as follows: 1 if <0.5 hours, 2 if 0.5-1 hours, 3 if 1-2 hours, 4 if 3-4 hours, 5 if 5-6 hours, 6 if 7-8 hours and 7 if 9-12 hours.
  The evening baseline measure was taken on the evening of Day -1 and the morning baseline measure was taken on the morning of Day 1 before cream was applied.
Time Frame: From baseline to Day 31
Population: Results were collected from a diary that participants were requested to fill in twice a day. Some participants missed some of the entries so there are less than 19 participants analysed for some of the time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Evening: Aprepitant 10 mg/g Gel; Morning: Aprepitant 10 mg/g Gel: 20 participants treated with aprepitant 10 mg/g gel on either left or right extremity
- Evening: Aprepitant Gel Vehicle; Morning: Aprepitant Gel Vehicle: 20 participants were treated with vehicle gel on either left or right extremity
Arm/Group | Evening: Aprepitant 10 mg/g Gel | Evening: Aprepitant Gel Vehicle | Morning: Aprepitant 10 mg/g Gel | Morning: Aprepitant Gel Vehicle
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  Day -1: number analyzed (Participants) | 15 | 15 | 19 | 19
  Day -1 | 3.7 (1.9) | 4.0 (2.1) | NA (NA) — Participants' assessments started on the evening of Day -1 so there is no morning data. | NA (NA) — Participants' assessments started on the evening of Day -1 so there is no morning data.
  Day 1: number analyzed (Participants) | 18 | 17 | 13 | 13
  Day 1 | 3.5 (1.7) | 3.7 (1.6) | 3.0 (1.8) | 3.4 (1.8)
  Day 2: number analyzed (Participants) | 19 | 18 | 19 | 19
  Day 2 | 3.0 (1.6) | 3.3 (1.7) | 3.2 (1.2) | 3.3 (1.3)
  Day 3 | 2.9 (1.4) | 3.3 (1.6) | 2.9 (1.1) | 3.1 (1.3)
  Day 4 | 2.7 (1.3) | 3.1 (1.4) | 2.8 (1.4) | 3.1 (1.5)
  Day 5: number analyzed (Participants) | 17 | 17 | 18 | 19
  Day 5 | 2.1 (1.2) | 2.7 (1.5) | 2.2 (1.2) | 2.8 (1.3)
  Day 6: number analyzed (Participants) | 18 | 19 | 18 | 19
  Day 6 | 2.5 (1.3) | 2.9 (1.4) | 2.3 (1.3) | 2.6 (1.5)
  Day 7: number analyzed (Participants) | 19 | 19 | 18 | 18
  Day 7 | 2.6 (1.3) | 2.9 (1.4) | 2.5 (1.5) | 2.7 (1.6)
  Day 8: number analyzed (Participants) | 18 | 18 | 19 | 18
  Day 8 | 2.4 (1.3) | 2.7 (1.5) | 2.3 (1.4) | 2.6 (1.5)
  Day 9: number analyzed (Participants) | 19 | 19 | 18 | 18
  Day 9 | 2.4 (1.3) | 2.8 (1.4) | 2.4 (1.3) | 2.8 (1.3)
  Day 10: number analyzed (Participants) | 19 | 18 | 18 | 19
  Day 10 | 2.4 (1.3) | 2.6 (1.5) | 2.4 (1.3) | 2.5 (1.4)
  Day 11: number analyzed (Participants) | 18 | 17 | 18 | 19
  Day 11 | 2.2 (1.4) | 2.8 (1.5) | 2.0 (1.3) | 2.4 (1.4)
  Day 12: number analyzed (Participants) | 17 | 17 | 18 | 18
  Day 12 | 2.1 (1.3) | 2.5 (1.4) | 2.2 (1.3) | 2.7 (1.3)
  Day 13: number analyzed (Participants) | 17 | 18 | 17 | 17
  Day 13 | 2.4 (1.6) | 2.7 (1.5) | 2.2 (1.5) | 2.5 (1.4)
  Day 14: number analyzed (Participants) | 19 | 19 | 18 | 19
  Day 14 | 2.1 (1.3) | 2.4 (1.4) | 2.1 (1.4) | 2.4 (1.3)
  Day 15: number analyzed (Participants) | 19 | 19 | 17 | 17
  Day 15 | 2.4 (1.4) | 2.5 (1.4) | 2.1 (1.5) | 2.5 (1.4)
  Day 16: number analyzed (Participants) | 19 | 19 | 16 | 17
  Day 16 | 2.2 (1.3) | 2.4 (1.4) | 2.1 (1.2) | 2.6 (1.2)
  Day 17: number analyzed (Participants) | 18 | 19 | 19 | 18
  Day 17 | 2.2 (1.3) | 2.5 (1.3) | 2.1 (1.4) | 2.6 (1.4)
  Day 18: number analyzed (Participants) | 18 | 19 | 18 | 19
  Day 18 | 2.1 (1.3) | 2.3 (1.2) | 2.2 (1.3) | 2.6 (1.3)
  Day 19: number analyzed (Participants) | 18 | 18 | 18 | 18
  Day 19 | 2.1 (1.3) | 2.4 (1.3) | 1.9 (1.3) | 2.3 (1.4)
  Day 20: number analyzed (Participants) | 18 | 19 | 16 | 18
  Day 20 | 2.0 (1.2) | 2.3 (1.2) | 2.0 (1.2) | 2.2 (1.2)
  Day 21: number analyzed (Participants) | 17 | 19 | 18 | 19
  Day 21 | 2.0 (1.3) | 2.2 (1.2) | 1.9 (1.3) | 2.1 (1.2)
  Day 22: number analyzed (Participants) | 17 | 17 | 17 | 19
  Day 22 | 1.9 (1.1) | 2.3 (1.2) | 2.0 (1.3) | 2.2 (1.2)
  Day 23: number analyzed (Participants) | 18 | 19 | 17 | 18
  Day 23 | 2.3 (1.5) | 2.4 (1.5) | 2.0 (1.2) | 2.3 (1.2)
  Day 24: number analyzed (Participants) | 17 | 15 | 17 | 17
  Day 24 | 1.9 (1.2) | 2.1 (1.2) | 2.0 (1.2) | 2.1 (1.2)
  Day 25: number analyzed (Participants) | 19 | 19 | 19 | 18
  Day 25 | 2.3 (1.4) | 2.5 (1.3) | 1.9 (1.2) | 2.1 (1.3)
  Day 26 | 2.2 (1.2) | 2.2 (1.3) | 2.4 (1.5) | 2.3 (1.5)
  Day 27: number analyzed (Participants) | 17 | 18 | 17 | 18
  Day 27 | 2.0 (1.2) | 2.1 (1.2) | 2.1 (1.2) | 2.2 (1.2)
  Day 28: number analyzed (Participants) | 8 | 8 | 18 | 19
  Day 28 | 1.8 (1.2) | 2.3 (1.2) | 2.0 (1.2) | 2.1 (1.2)
  Day 29: number analyzed (Participants) | 2 | 2 | 6 | 6
  Day 29 | 1.0 (0.0) | 2.0 (0.0) | 1.5 (1.2) | 1.7 (1.2)
  Day 30: number analyzed (Participants) | 1 | 1 | 2 | 2
  Day 30 | 1.0 (NA) — This value has not been calculated because only one person was analyzed. | 2.0 (NA) — This value has not been calculated because only one person was analyzed. | 1.0 (0.0) | 1.5 (0.7)
  Day 31: number analyzed (Participants) | 19 | 19 | 1 | 1
  Day 31 | NA (NA) — Participants' assessments ended on the morning of Day 31 so there is no evening data. | NA (NA) — Participants' assessments ended on the morning of Day 31 so there is no evening data. | 1.0 (NA) — This value has not been calculated because only one person was analyzed. | 2.0 (NA) — This value has not been calculated because only one person was analyzed.

14. Secondary Outcome: Daily Assessments of Average Pruritus by Use of a VAS
Description: During the trial participants completed a diary twice daily, in the morning and in the evening, each covering the preceding 12 hours, which collected the average intensity of pruritus since last evaluation by use of a VAS (ranging from 0 to 100). The participants assessed the intensity of present pruritus of each treated area on a visual analogue scale (VAS) with a score of "0" (no itch at all) to "10" (worst imaginable itch) at the two extremes on a 100 mm line.
  The evening baseline measure was taken on the evening of Day -1 and the morning baseline measure was taken on the morning of Day 1, before cream was applied.
Time Frame: From baseline to Day 31
Population: Results were collected from a diary that participants were requested to fill in twice a day. Some participants missed some of the entries so there are less than 20 participants analysed for some of the time points.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Evening: Aprepitant 10 mg/g Gel | Evening: Aprepitant Gel Vehicle | Morning: Aprepitant 10 mg/g Gel | Morning: Aprepitant Gel Vehicle
Number analyzed (Participants) | 20 | 20 | 20 | 20
mm
  Day -1: number analyzed (Participants) | 15 | 15 | 20 | 20
  Day -1 | 49.1 (20.9) | 51.3 (21.1) | NA (NA) — Participants' assessments started on the evening of Day -1 so there is no morning data. | NA (NA) — Participants' assessments started on the evening of Day -1 so there is no morning data.
  Day 1: number analyzed (Participants) | 18 | 19 | 14 | 14
  Day 1 | 45.0 (21.5) | 44.7 (21.7) | 46.9 (21.6) | 49.3 (20.6)
  Day 2: number analyzed (Participants) | 19 | 18 | 20 | 20
  Day 2 | 35.1 (24.1) | 38.9 (22.2) | 38.3 (18.4) | 39.2 (19.0)
  Day 3: number analyzed (Participants) | 20 | 20 | 19 | 19
  Day 3 | 33.7 (21.0) | 35.8 (20.4) | 33.6 (21.0) | 33.7 (19.7)
  Day 4: number analyzed (Participants) | 19 | 19 | 20 | 20
  Day 4 | 31.8 (20.2) | 37.5 (18.3) | 34.5 (22.1) | 37.2 (18.7)
  Day 5: number analyzed (Participants) | 18 | 18 | 19 | 19
  Day 5 | 27.4 (19.6) | 31.0 (18.0) | 24.2 (16.3) | 33.7 (16.9)
  Day 6: number analyzed (Participants) | 18 | 19 | 19 | 20
  Day 6 | 26.4 (15.9) | 31.5 (17.6) | 26.8 (17.4) | 30.3 (19.1)
  Day 7: number analyzed (Participants) | 20 | 20 | 18 | 18
  Day 7 | 30.4 (21.7) | 33.2 (22.2) | 28.3 (20.9) | 31.9 (21.9)
  Day 8: number analyzed (Participants) | 18 | 18 | 20 | 19
  Day 8 | 23.3 (12.6) | 28.8 (16.1) | 26.5 (18.4) | 30.1 (18.8)
  Day 9: number analyzed (Participants) | 20 | 20 | 18 | 18
  Day 9 | 24.5 (16.6) | 27.6 (17.9) | 26.8 (17.1) | 27.4 (16.0)
  Day 10: number analyzed (Participants) | 19 | 18 | 19 | 20
  Day 10 | 22.0 (14.8) | 28.2 (17.7) | 30.6 (21.6) | 30.2 (20.6)
  Day 11: number analyzed (Participants) | 19 | 19 | 18 | 19
  Day 11 | 23.3 (18.8) | 28.4 (19.1) | 22.3 (15.2) | 29.3 (19.0)
  Day 12: number analyzed (Participants) | 17 | 17 | 19 | 19
  Day 12 | 19.9 (13.4) | 23.7 (12.6) | 23.0 (17.0) | 27.8 (16.8)
  Day 13: number analyzed (Participants) | 19 | 19 | 18 | 18
  Day 13 | 21.8 (26.0) | 26.4 (14.8) | 20.2 (13.4) | 23.4 (14.5)
  Day 14: number analyzed (Participants) | 20 | 20 | 19 | 19
  Day 14 | 20.9 (15.4) | 23.1 (13.7) | 21.9 (15.1) | 24.7 (16.1)
  Day 15: number analyzed (Participants) | 19 | 20 | 17 | 17
  Day 15 | 24.2 (16.9) | 25.2 (16.0) | 19.3 (14.6) | 22.1 (13.0)
  Day 16: number analyzed (Participants) | 19 | 20 | 18 | 19
  Day 16 | 20.8 (13.6) | 24.3 (16.7) | 22.7 (15.4) | 25.4 (15.3)
  Day 17: number analyzed (Participants) | 19 | 19 | 20 | 19
  Day 17 | 20.2 (14.6) | 21.7 (14.8) | 18.8 (14.4) | 22.8 (14.3)
  Day 18: number analyzed (Participants) | 19 | 20 | 19 | 20
  Day 18 | 18.5 (13.6) | 21.1 (14.5) | 21.6 (13.9) | 22.8 (13.0)
  Day 19: number analyzed (Participants) | 19 | 19 | 19 | 19
  Day 19 | 15.6 (11.2) | 19.9 (16.0) | 20.7 (14.9) | 22.4 (14.7)
  Day 20: number analyzed (Participants) | 19 | 20 | 18 | 20
  Day 20 | 16.0 (11.9) | 19.7 (12.9) | 17.8 (13.1) | 18.6 (14.9)
  Day 21: number analyzed (Participants) | 18 | 20 | 19 | 20
  Day 21 | 14.5 (14.6) | 17.0 (16.4) | 16.1 (13.2) | 17.1 (12.4)
  Day 22: number analyzed (Participants) | 18 | 19 | 19 | 20
  Day 22 | 14.3 (13.2) | 15.9 (15.1) | 15.3 (14.4) | 16.6 (12.8)
  Day 23: number analyzed (Participants) | 20 | 20 | 19 | 20
  Day 23 | 15.6 (13.6) | 17.2 (14.3) | 15.8 (16.0) | 14.6 (12.7)
  Day 24: number analyzed (Participants) | 17 | 17 | 19 | 19
  Day 24 | 15.7 (14.1) | 16.7 (15.1) | 16.5 (16.6) | 15.5 (13.4)
  Day 25 | 18.2 (16.4) | 16.8 (14.0) | 15.8 (14.8) | 16.5 (17.0)
  Day 26: number analyzed (Participants) | 19 | 20 | 20 | 20
  Day 26 | 15.1 (13.1) | 16.6 (15.8) | 19.8 (17.3) | 16.3 (13.5)
  Day 27: number analyzed (Participants) | 19 | 19 | 20 | 20
  Day 27 | 14.2 (15.4) | 14.1 (12.9) | 13.6 (13.8) | 14.6 (13.0)
  Day 28: number analyzed (Participants) | 8 | 8 | 19 | 20
  Day 28 | 7.8 (7.5) | 11.6 (10.6) | 16.4 (14.5) | 14.9 (13.5)
  Day 29: number analyzed (Participants) | 20 | 20 | 7 | 7
  Day 29 | 3.0 (2.8) | 5.5 (2.1) | 4.7 (6.1) | 4.9 (5.6)
  Day 30: number analyzed (Participants) | 1 | 1 | 2 | 2
  Day 30 | 3.0 (NA) — This value has not been calculated because only one person was analyzed. | 3.0 (NA) — This value has not been calculated because only one person was analyzed. | 3.5 (2.1) | 3.5 (0.7)
  Day 31: number analyzed (Participants) | 1 | 1 | 1 | 1
  Day 31 | NA (NA) — Participants' assessments ended on the morning of Day 31 so there is no evening data. | NA (NA) — Participants' assessments ended on the morning of Day 31 so there is no evening data. | 2.0 (NA) — This value has not been calculated because only one person was analyzed. | 2.0 (NA) — This value has not been calculated because only one person was analyzed.

15. Secondary Outcome: Daily Assessments of Maximum Intensity of Pruritus by Use of a VAS
Description: During the trial participants completed a diary twice daily, in the morning and in the evening, each covering the preceding 12 hours, which collected the maximum intensity of pruritus since last evaluation by use of a VAS (ranging from 0 to 100). The participants assessed the intensity of present pruritus of each treated area on a visual analogue scale (VAS) with a score of "0" (no itch at all) to "10" (worst imaginable itch) at the two extremes on a 100 mm line.
  The evening baseline measure was taken on the evening of Day -1 and the morning baseline measure was taken on the morning of Day 1 before cream was applied.
Time Frame: From baseline to Day 31
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Evening: Aprepitant 10 mg/g Gel; Evening: Aprepitant Gel Vehicle; Morning: Aprepitant Gel Vehicle: 20 participants were treated with vehicle gel on either left or right extremity
Arm/Group | Evening: Aprepitant 10 mg/g Gel | Evening: Aprepitant Gel Vehicle | Morning: Aprepitant 10 mg/g Gel | Morning: Aprepitant Gel Vehicle
Number analyzed (Participants) | 20 | 20 | 20 | 20
mm
  Day -1: number analyzed (Participants) | 15 | 15 | 20 | 20
  Day -1 | 61.1 (21.8) | 62.7 (25.7) | NA (NA) — Participants' assessments started on the evening of Day -1 so there is no morning data. | NA (NA) — Participants' assessments started on the evening of Day -1 so there is no morning data.
  Day 1: number analyzed (Participants) | 19 | 18 | 14 | 14
  Day 1 | 49.9 (25.4) | 54.7 (24.6) | 56.0 (25.3) | 62.4 (22.0)
  Day 2: number analyzed (Participants) | 19 | 18 | 20 | 20
  Day 2 | 43.2 (24.7) | 46.7 (25.1) | 48.8 (22.2) | 46.7 (23.0)
  Day 3: number analyzed (Participants) | 20 | 20 | 19 | 19
  Day 3 | 41.6 (24.7) | 42.7 (24.8) | 39.5 (24.5) | 43.6 (23.5)
  Day 4: number analyzed (Participants) | 19 | 19 | 20 | 20
  Day 4 | 37.7 (21.7) | 42.8 (19.9) | 39.5 (25.1) | 47.7 (20.7)
  Day 5: number analyzed (Participants) | 18 | 18 | 19 | 19
  Day 5 | 33.4 (23.4) | 39.7 (23.6) | 32.3 (20.1) | 41.7 (21.9)
  Day 6: number analyzed (Participants) | 18 | 19 | 19 | 20
  Day 6 | 34.1 (19.5) | 38.4 (21.0) | 34.3 (21.1) | 39.1 (24.5)
  Day 7: number analyzed (Participants) | 20 | 20 | 18 | 18
  Day 7 | 35.2 (23.5) | 39.2 (24.2) | 35.3 (23.5) | 38.9 (24.5)
  Day 8: number analyzed (Participants) | 18 | 18 | 20 | 19
  Day 8 | 31.4 (16.1) | 37.4 (19.5) | 32.2 (20.3) | 40.7 (23.0)
  Day 9: number analyzed (Participants) | 20 | 20 | 18 | 18
  Day 9 | 32.0 (20.0) | 35.0 (21.5) | 32.8 (18.8) | 35.9 (18.5)
  Day 10: number analyzed (Participants) | 19 | 18 | 19 | 20
  Day 10 | 29.4 (18.0) | 34.5 (19.7) | 40.0 (22.8) | 41.1 (22.5)
  Day 11: number analyzed (Participants) | 19 | 19 | 18 | 19
  Day 11 | 30.7 (22.4) | 37.3 (23.0) | 28.7 (17.8) | 36.8 (21.1)
  Day 12: number analyzed (Participants) | 17 | 17 | 19 | 19
  Day 12 | 27.1 (17.2) | 31.8 (16.8) | 31.6 (22.8) | 38.6 (20.8)
  Day 13: number analyzed (Participants) | 19 | 19 | 18 | 18
  Day 13 | 31.0 (21.9) | 34.2 (21.8) | 29.1 (21.7) | 31.3 (21.3)
  Day 14: number analyzed (Participants) | 20 | 20 | 19 | 20
  Day 14 | 27.1 (19.6) | 31.2 (19.0) | 30.7 (21.2) | 31.9 (21.7)
  Day 15: number analyzed (Participants) | 20 | 20 | 17 | 17
  Day 15 | 29.4 (19.0) | 32.1 (18.9) | 26.3 (19.1) | 30.7 (19.3)
  Day 16: number analyzed (Participants) | 19 | 20 | 18 | 19
  Day 16 | 28.2 (16.8) | 32.8 (18.3) | 29.1 (18.9) | 32.9 (19.5)
  Day 17: number analyzed (Participants) | 19 | 20 | 20 | 20
  Day 17 | 28.2 (19.1) | 29.3 (21.8) | 25.5 (16.7) | 29.8 (17.1)
  Day 18: number analyzed (Participants) | 19 | 20 | 19 | 20
  Day 18 | 25.6 (16.2) | 27.7 (17.1) | 29.2 (18.5) | 30.4 (16.8)
  Day 19: number analyzed (Participants) | 19 | 19 | 19 | 19
  Day 19 | 24.1 (15.7) | 27.4 (19.8) | 27.7 (20.2) | 33.1 (21.7)
  Day 20: number analyzed (Participants) | 19 | 20 | 18 | 20
  Day 20 | 25.1 (17.4) | 27.1 (18.0) | 23.2 (14.5) | 23.5 (17.6)
  Day 21: number analyzed (Participants) | 18 | 20 | 19 | 20
  Day 21 | 21.3 (19.5) | 23.0 (19.0) | 22.6 (16.2) | 25.7 (19.7)
  Day 22: number analyzed (Participants) | 18 | 19 | 19 | 20
  Day 22 | 20.8 (19.5) | 21.5 (16.7) | 20.1 (16.8) | 22.7 (15.1)
  Day 23: number analyzed (Participants) | 20 | 20 | 19 | 20
  Day 23 | 22.2 (17.9) | 24.2 (18.0) | 23.2 (22.3) | 21.1 (16.7)
  Day 24: number analyzed (Participants) | 17 | 17 | 18 | 19
  Day 24 | 21.1 (18.4) | 22.0 (19.1) | 20.8 (17.5) | 21.1 (16.6)
  Day 25 | 22.7 (19.3) | 23.8 (21.3) | 21.8 (20.1) | 20.8 (17.3)
  Day 26: number analyzed (Participants) | 19 | 20 | 20 | 20
  Day 26 | 23.2 (18.4) | 24.0 (19.2) | 24.1 (20.2) | 23.1 (18.7)
  Day 27: number analyzed (Participants) | 19 | 19 | 20 | 20
  Day 27 | 20.9 (21.8) | 23.1 (21.3) | 19.6 (18.6) | 21.3 (18.8)
  Day 28: number analyzed (Participants) | 8 | 8 | 19 | 20
  Day 28 | 12.6 (11.9) | 18.9 (20.1) | 24.7 (19.9) | 24.7 (21.7)
  Day 29: number analyzed (Participants) | 2 | 2 | 7 | 7
  Day 29 | 3.5 (2.1) | 7.5 (0.7) | 5.7 (7.0) | 5.9 (4.3)
  Day 30: number analyzed (Participants) | 1 | 1 | 2 | 2
  Day 30 | 2.0 (NA) — This value has not been calculated because only one person was analyzed. | 4.0 (NA) — This value has not been calculated because only one person was analyzed. | 4.5 (0.7) | 5.5 (0.7)
  Day 31: number analyzed (Participants) | 20 | 20 | 1 | 1
  Day 31 | NA (NA) — Participants' assessments ended on the morning of Day 31 so there is no evening data. | NA (NA) — Participants' assessments ended on the morning of Day 31 so there is no evening data. | 3.0 (NA) — This value has not been calculated because only one person was analyzed. | 4.0 (NA) — This value has not been calculated because only one person was analyzed.

16. Secondary Outcome: Percent Change From Baseline in Pruritis Assessed by VAS at End of Treatment
Description: On the last day of treatment, participants assessed the change of pruritus compared to baseline in percentage by use of a VAS (ranging from 0 to 100). The participants assessed the intensity of present pruritus of each treated area on a visual analogue scale (VAS) with a score of "0" (no itch at all) to "10" (worst imaginable itch) at the two extremes on a 100 mm line.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Aprepitant 10 mg/g Gel | Aprepitant Gel Vehicle
Number analyzed (Participants) | 20 | 20
percent change | 50.8 (28.1) | 41.7 (29.2)

ADVERSE EVENTS:
Time Frame: From Day 1 to Day 42
Groups:
- Treatment Not Defined: The treatment for these adverse events are not defined
- Aprepitant Gel Vehicle: Placebo (Aprepitant gel vehicle)
- Aprepitant Gel: 10 mg/g aprepitant gel
Arm/Group | Treatment Not Defined | Aprepitant Gel Vehicle | Aprepitant Gel
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 10/20 | 15/20 | 11/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Not Defined (N=20) | Aprepitant Gel Vehicle (N=20) | Aprepitant Gel (N=20)
Visual impairment (Eye disorders) | 1 | 0 | 0
Application site discolouration (General disorders) | 0 | 0 | 1
Application site discomfort (General disorders) | 0 | 2 | 4
Application site erythema (General disorders) | 0 | 1 | 1
Application site haemorrhage (General disorders) | 0 | 1 | 0
Application site nodule (General disorders) | 0 | 1 | 1
Application site pain (General disorders) | 0 | 11 | 8
Application site paraesthesia (General disorders) | 0 | 2 | 1
Application site pruritus (General disorders) | 0 | 1 | 1
Application site urticaria (General disorders) | 0 | 1 | 2
Application site vesicles (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Wound treatment (Surgical and medical procedures) | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting or presenting a manuscript relating to the clinical trial to a publisher, reviewer or other outside person, the Investigator shall submit to LEO, in writing, a copy of the intended publication, describing the detail of any Research Results that the Investigator intends to Publish, at least 60 days before the date of the proposed submission for publication.